CLINICAL TRIAL: NCT03293147
Title: BiOmarkers in Urine, anTihypeRtensive trEAtment and Blood Pressure Control in Hypertensive Patients
Brief Title: OUTREACH: Urine Analysis and Antihypertensive Treatment
Acronym: OUTREACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: British Heart Foundation (Other); Manchester Academic Health Science Centre (Other); Omron Healthcare Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Maciej Tomaszewski, Professor of Cardiovascular Medicine, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R120993
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Hypertension; Adherence, Medication
Keywords: Blood pressure; Antihypertensive treatment; Adherence; Biomarker; Urine; HPLC-MS/MS
MeSH Terms: conditions — Hypertension; Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Multi-center randomised controlled trial
Who Masked: Participant, Investigator
Masking Description: Participants and clinicians will initially be blinded to the result of the baseline (at trial entry) HPLC-MS/MS based urine test to determine the participant adherence to antihypertensive treatment.
  Non-adherent patients allocated to Arm A will be un-blinded at the stage of visit 3 where the results of their HPLC-MS/MS urine test will be revealed to them as a part of HPLC-MS/MS-guided intervention. The doctor will also require un-blinding to provide the required intervention. However, during further study visits the research personnel will remain blinded as to the adherence status of these patients, the results of their HPLC-MS/MS-based analysis and the treatment allocation. The doctor who delivers the intervention will not be involved in collecting clinical information necessary to define outcomes during appointments 4 and 5.
  Hypertensive patients randomised to Arms B and C will remain blinded to the results of their HPLC-MS/MS-based urine test throughout all stages of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Intervention group: Non-adherent hypertensive patients randomised in Arm A will receive standard clinical care plus HPLC-MS/MS-guided intervention.
  Interventions: Other: HPLC-MS/MS-guided intervention
- Arm B (Active Comparator): Control group: Non-adherent hypertensive patients randomised in Arm B will receive clinical standard care.
  Interventions: Other: Standard care
- Arm C (Active Comparator): Control group: Adherent hypertensive patients randomised in Arm C will receive clinical standard care.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: HPLC-MS/MS-guided intervention — The HPLC-MS/MS-guided intervention consists of providing partially or totally non-adherent hypertensive patients with information on the results of their HPLC-MS/MS-based urine analysis combined with tailored targeting of the main reason(s) for the deviation from the prescribed antihypertensive treatment
  Arms: Arm A
Other: Standard care — Standard care for hypertensive patients
  Arms: Arm B; Arm C

SUMMARY:
Non-adherence to antihypertensive treatment is one of the leading causes of suboptimal blood pressure control and translates into increased risk of cardiovascular morbidity and mortality. Currently, there is no effective intervention for therapeutic non-adherence. Our project will assess whether high performance liquid chromatography mass spectrometry (HPLC-MS/MS)-guided intervention (providing patients with information on the results of their HPLC-MS/MS-based urine analysis combined with targeting the main reason for non-adherence) leads to an improvement in blood pressure control, adherence and a reduction in healthcare costs. Our multicentre prospective randomised controlled trial consists of 6 stages (screening, recruitment, baseline phenotype assessment, intervention, short-term and long-term outcome visits). The study will fill in an important gap in knowledge on management of blood pressure in non-adherent hypertensive patients beyond the initial diagnostic step. It will also inform the development of a cost-effective model for the management of non-adherence in chronic disorders that require long-term drug therapy.

DETAILED DESCRIPTION:
Non-adherence to antihypertensive treatment is one of the leading causes of suboptimal blood pressure control and translates into increased risk of cardiovascular morbidity and mortality. Currently, there is no effective intervention for therapeutic non-adherence.

An ultra-sensitive and highly specific biochemical assay has been developed to detect urinary biomarkers of antihypertensive treatment. The high performance liquid chromatography mass spectrometry (HPLC-MS/MS)-based assay screens spot urine samples for the presence of 40 commonly prescribed blood pressure lowering medications. The results of the test provide a clinician with information on the presence/absence of prescribed antihypertensive drugs or/and their metabolites in urine - a direct confirmation of therapeutic adherence/non-adherence.

The study is a prospective multi-centre randomised controlled trial to examine if HPLC-MS/MS-guided intervention is superior to standard clinical care in improving clinical, behavioural and health-economy outcomes in hypertensive patients who are non-adherent to antihypertensive treatment.

Patient adherence to antihypertensive treatment will be determined at baseline. Non-adherent hypertensive patients at baseline will be randomised in a 1:1 ration to either usual clinical care plus HPLC-MS/MS-guided intervention (Arm A) or usual clinical care only (Arm B).

The study also evaluates a cohort of patients who are adherent to antihypertensive treatment at baseline. Those adherent hypertensive patients will receive the usual clinical care (Arm C). The main purpose of involving this group of patients is to blind the clinical research staff to the adherence status of those patients randomised receiving standard care alone, to prevent introducing any bias in treating non-adherent patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or above
* Patients previously diagnosed with and pharmacologically managed for hypertension
* Patients with antihypertensive treatment with at least two antihypertensive medications
* Patients have full capability of providing informed consent

Exclusion Criteria:

* Patients with recent history of admission to the hospital relating to their hypertension or treatment with anti-hypertensive medications (<2 weeks) (i)
* Patient refusal for 7-day home-based blood pressure monitoring (7-HBBPM)
* Self-reported pregnancy or breastfeeding
* Female patients planning to conceive within the next 6 months

  (i) Including admission to A&E

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Clinic systolic blood pressure | visit 4 (short term follow-up; approx. 3 months post intervention, when feasible to conduct)
  Blood pressure measurements will be taken after 5 minutes of rest in a sitting position with an electronic digital Omron monitor and the cuff size adjusted to the arm circumference as per international guidelines. Three measurements of systolic blood pressure will be taken in a row (separated by approximately 1 minute interval) and recorded at every visit

SECONDARY OUTCOMES:
Change in clinic systolic blood pressure | visit 5 (long term follow-up; ~4.5 months post intervention, when feasible to conduct)
  Blood pressure measurements will be taken after 5 minutes of rest in a sitting position with an electronic digital Omron monitor and the cuff size adjusted to the arm circumference as per international guidelines. Three measurements of systolic blood pressure will be taken in a row (separated by approximately 1 minute interval) and recorded at every visit
Change in clinic diastolic blood pressure | visit 4 (short term follow-up; ~3 months post intervention, when feasible to conduct)
  Blood pressure measurements will be taken after 5 minutes of rest in a sitting position with an electronic digital Omron monitor and the cuff size adjusted to the arm circumference as per international guidelines. Three measurements of diastolic blood pressure will be taken in a row (separated by approximately 1 minute interval) and recorded at every visit
Change in clinic diastolic blood pressure | visit 5 (long term follow-up; ~4.5 months post intervention, when feasible to conduct)
  Blood pressure measurements will be taken after 5 minutes of rest in a sitting position with an electronic digital Omron monitor and the cuff size adjusted to the arm circumference as per international guidelines. Three measurements of diastolic blood pressure will be taken in a row (separated by approximately 1 minute interval) and recorded at every visit
Change in home blood pressure | visit 4 (short term follow-up; ~3 months post intervention, when feasible to conduct)
  This measurement will be conducted using oscillometric Omron monitors. Patients will be handed the monitors by the research nurses at each visit and will be provided instructions to use the Omron monitor. While all blood pressure measurements will be stored automatically on the monitors, patients will be also asked to keep a written record on paper (to avoid loss of data in case a monitor stops working or goes out of order).
Change in home blood pressure | visit 5 (long term follow-up; ~4.5 months post intervention, when feasible to conduct)
  This measurement will be conducted using oscillometric Omron monitors. Patients will be handed the monitors by the research nurses at each visit and will be provided instructions to use the Omron monitor. While all blood pressure measurements will be stored automatically on the monitors, patients will be also asked to keep a written record on paper (to avoid loss of data in case a monitor stops working or goes out of order).
Change in biochemical adherence of patients | visit 2 (~3 weeks post recruitment, when feasible to conduct)
  HPLC-MS/MS test will determine the numbers and list of antihypertensive drugs detected in the patient urine sample and this will be compared to the patient prescription
Change in biochemical adherence of patients | visit 4 (short term follow-up; ~3 months post intervention, when feasible to conduct)
  HPLC-MS/MS test will determine the numbers and list of antihypertensive drugs detected in the patient urine sample and this will be compared to the patient prescription.
Change in biochemical adherence of patients | visit 5 (long term follow-up; ~4.5 months post intervention, when feasible to conduct)
  HPLC-MS/MS test will determine the numbers and list of antihypertensive drugs detected in the patient urine sample and this will be compared to the patient prescription.
Change in urinary albumin / creatinine ratio | visit 4 (short term follow-up; ~3 months post intervention, when feasible to conduct)
  Urinary albumin / creatinine ratio is a urinary marker of target organ damage.
Change in urinary albumin / creatinine ratio | visit 5 (long term follow-up; ~4.5 months post intervention, when feasible to conduct)
  Urinary albumin / creatinine ratio is a urinary marker of target organ damage.
Changes in health economy parameters | visit 4 (short term follow-up; ~3 months post intervention, when feasible to conduct)
  Health economy parameters (collected via questionnaires) will be calculated over the study time horizon to determine total costs of clinical/social care
Changes in health economy parameters | visit 5 (long term follow-up; ~4.5 months post intervention, when feasible to conduct)
  Health economy parameters (collected via questionnaires) will be calculated over the study time horizon to determine total costs of clinical/social care

OTHER OUTCOMES:
Changes in psychological profile | visit 4 (short term follow-up; ~3 months post intervention, when feasible to conduct)
  Psychological questionnaires assessing participants perspectives of treatment will be completed by patient when attending clinic visit 1, 4 and 5
Changes in psychological profile | visit 5 (long term follow-up; ~4.5 months post intervention, when feasible to conduct)
  Psychological questionnaires assessing participants perspectives of treatment will be completed by patient when attending clinic visit 1, 4 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Tomaszewski, Prof., MD, Principal Investigator — University of Manchester
Locations (12):
- United Kingdom (12):
  - University College London Hospitals NHS Foundation Trust, London, Greater London
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - Ninewells Hospital, Dundee, Scotland
  - Alvaston Medical Centre, Derby
  - Epsom & St. Helier University Hospitals NHS Trust, Epsom
  - Glenfield General Hospital, Leicester
  - Royal Free Hospital, London
  - Guy's and St Thomas' Hospital, London
  - Homerton Hospital, London
  - St Bartholomews Hospital, London
  - Chilwell Valley and Meadows Practice, Nottingham
  - University Hospitals Dorset NHS Foundation Trust, Poole

IPD SHARING:
Plan to Share IPD: No